CLINICAL TRIAL: NCT03581435
Title: A Study of Circulating Exosome Proteomics In Gallbladder Carcinoma Patients
Acronym: EXOGBC001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: liu yingbin (Other)
Collaborators: The First Hospital of Jilin University (Other); Shanghai Zhongshan Hosiptal (Unknown); The First Affiliated Hospital of Bengbu Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Jining Medical University (Other); The Affiliated Hospital of Tianjin Medical University (Unknown); The first affiliated hospital of Zhongshan university (Unknown)
Responsible Party: Sponsor-Investigator, liu yingbin, vice-president，Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: EXOGBC001
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Proteinosis; Gallbladder Carcinoma
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gallbladder carcinoma patients: Cases will be the patients with newly-diagnosed gallbladder carcinoma.
- The controls: The controls will be matched （1：1）by sex，race and age which will be selected from the patients receiving cholecystectomy due to gallstones from the same hospital with the cases.

SUMMARY:
This research will be the first study for exosome purified from blood in gallbladder carcinoma patients. Proteomics studies will be done in both tumor tissue and the circulating exosome from blood specimens. Then, the potential prognostic and predictive biomarkers will be searched by bioinformatics to find the correlations between exosome biomarkers and gallbladder carcinoma.

DETAILED DESCRIPTION:
Background:

Exosomes are formed by inward budding of late endosomes, producing multivesicular bodies (MVBs), and are released into the environment by fusion of the MVBs with the plasma membrane. It has been demonstrated that the content and function of exosomes depends on the originating cell and the conditions under which they are produced. Tumor exosome production, transfer and education of bone marrow cells supports tumor growth and metastasis.

Aims of the study:

Proteomics studies will be done in both tumor tissue and the circulating exosome from the gallbladder carcinoma patients. Then, the potential prognostic and predictive biomarkers will be searched by bioinformatics to find the correlations between exosome biomarkers and gallbladder carcinoma.

Materials and Methods:

The investigators will conduct a case-control study in 11 hospitals from China. Cases will be the patients with newly-diagnosed gallbladder carcinoma. The controls will be matched （1：1）by sex，race and age which will be selected from the patients receiving cholecystectomy due to gallstones from the same hospital with the cases. A total of 50 patients with gallbladder carcinoma will be recruited. The investigators will obtain the blood and tumor tissue samples for further analysis of proteomics studies. Exosome from blood specimens will be isolated and purified by sucrose gradient ultracentrifugation. The potential prognostic and predictive biomarkers will be searched by bioinformatics to find the correlations between exosome biomarkers and gallbladder carcinoma. Data will be collected from January 2018 to December 2018.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gallbladder carcinoma by imaging tests (cases) Diagnosed with chronic cholecystitis by imaging tests (hospital controls)

Exclusion Criteria:

* The pathology diagnosis and imaging does not matched Patients with other malignant tumors Patients with other severe systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will conduct a case-control study in 11 hospitals from China. Cases will be the patients with newly-diagnosed gallbladder carcinoma. The controls will be matched （1：1）by sex，race and age which will be selected from the patients receiving cholecystectomy due to gallstones from the same hospital with the cases. A total of 50 patients with gallbladder carcinoma will be recruited.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the protein profile in tumor derived exosomes from the gallbladder carcinoma patients | Up to 2 years from start of study
  Proteomics studies will be done in both tumor tissue and the circulating exosomes from blood specimens. The specific protein A in the circulating exosomes from the gallbladder carcinoma patients will be selected for further analysis.
The expression of protein A in the circulating exosomes from patients | Up to 2 years from start of study
  The expression of protein A （which is selected from outcome 1） in the circulating exosomes from patients will be detected by flow cytometry analysis. The ROC curve of A+ circulating exosomes will be done to compare with the clinical standard tumour biomarker (e.g. CA199) for patients with gallbladder carcinoma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China